CLINICAL TRIAL: NCT07353346
Title: Evaluation of Short-term and Long-term Efficacy of Endoscopic Treatment for Gastrointestinal Submucosal Tumors
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJLL-KY-20252474
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Submucosal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to comprehensively assess how well endoscopic treatments work for gastrointestinal submucosal tumors (SMTs)-both in the short term right after treatment and over the long run-and to figure out what factors might affect the treatment's success. Specifically, it seeks to answer key questions: How effective are common endoscopic procedures at removing these tumors completely? What are the risks of complications like bleeding or perforation after treatment? Do patients stay healthy without the tumor coming back in the years following treatment? And what aspects (such as tumor size, location, or the type of endoscopic method used) influence whether the treatment works well or leads to problems? Study Description and Hypothesis Gastrointestinal submucosal tumors are growths that develop beneath the inner lining of the digestive tract (like the esophagus, stomach, or intestines). Unlike traditional open surgery, endoscopic treatments are minimally invasive-doctors use thin, flexible tubes with cameras and tools to remove tumors through natural body openings, which typically means smaller wounds, faster recovery, and no visible scars. However, there's still limited clear information about how well these treatments hold up over time or which patients benefit most.

This study is a retrospective analysis, meaning researchers will look back at the medical records of 700 patients who received endoscopic treatment for SMTs at Xijing Hospital between January 2012 and August 2025. The team will collect details like the tumor's size and location, the specific endoscopic method used (such as EMR, ESE, STER, or EFR), how long the procedure took, whether any complications occurred, and follow-up results to check for recurrence.

The study's core hypothesis is that endoscopic treatments are safe and effective for gastrointestinal submucosal tumors-successfully removing most tumors with low complication rates-and that factors like the tumor's size, where it's located in the digestive tract, and the type of endoscopic technique used will play a role in how well the treatment works and whether the tumor comes back later. By analyzing these past cases, the research hopes to provide reliable information to help doctors choose the best treatment for patients with SMTs in the future, ensuring more personalized and effective care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent endoscopic treatment for gastrointestinal submucosal tumors at Xijing Hospital from January 1, 2012 to August 1, 2025.

Exclusion Criteria:

* Patients with gastrointestinal protruding lesions caused by external compression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent endoscopic treatment for gastrointestinal submucosal tumors at Xijing Hospital from January 1, 2012 to August 1, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Surgical success rate | Three days after the operation
  The surgical success rate is defined as the operation completion rate
long-term prognosis of patients | Taking 1 year, 3 years, and 5 years after surgery
  long-term prognosis concerns the disease progression at 1 year, 3 years, and 5 years after surgery.